CLINICAL TRIAL: NCT04999696
Title: Minimally Invasive Therapy Versus Open Radical Hysterectomy (MITOR) for Management of Early Stage Cervical Cancer
Brief Title: Minimally Invasive Therapy Versus Open Radical Hysterectomy for Management of Early Stage Cervical Cancer
Acronym: MITOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201902269A3
Record Dates: First submitted 2021-07-12; First posted 2021-08-11 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2022-07

CONDITIONS: Cancer of Cervix; Laparoscopic Surgery
Keywords: Cervical cancer; Radical hysterectomy; Laparotomy; Laparoscopy; Outcome
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic radical hysterectomy (Experimental)
  Interventions: Procedure: radical hysterectomy
- Laparotomic radical hysterectomy (Active Comparator)
  Interventions: Procedure: radical hysterectomy

INTERVENTIONS:
Procedure: radical hysterectomy — To compare disease-free survival and overall survival of patients with early stage cervical cancer undergoing total laparoscopic radical hysterectomy versus total abdominal radical hysterectomy

SUMMARY:
Radical hysterectomy and pelvic lymph node dissection (+/- aortic lymph node dissection) is the standard treatment for early stage cervical cancer. And minimally invasive surgery has been successfully and safely demonstrated in the treatment of early stage cervical cancer. This study aims to compare total laparoscopic radical hysterectomy and total abdominal radical hysterectomy in terms of disease-free survival and overall survival. Rates and characteristics of recurrence, incidence of complications and morbidity, impact on quality of life and cost-effectiveness will also be determined.

DETAILED DESCRIPTION:
Radical hysterectomy and pelvic lymph node dissection (+/- aortic lymph node dissection) is the standard treatment for early stage cervical cancer. Laparotomy has been the surgical method of choice for a considerable length of time. While it is an accepted effective treatment, laparotomy is highly invasive and is associated with increased risk of tissue trauma, intraoperative and postoperative complications, and longer hospital stay.

Minimally invasive surgery has been successfully and safely demonstrated in the treatment of early stage cervical cancer. Retrospective studies have shown that oncologic outcomes in terms of recurrence rates and patterns of recurrence are similar in patients who had a laparoscopic or an open approach to radical hysterectomy. There is reduction of overall postoperative complications, treatment-related morbidity and length of hospital stay. However, there are two studies stating poorer survival of women treated by minimally invasive surgery. An epidemiologic study using two large US databases (National Cancer Database and Surveillance, Epidemiology, and End Results database) showed a reduction in overall survival of patients undergoing minimally invasive radical hysterectomy. Furthermore, in a prospective, multi-center, open-label randomized clinical trial, minimally invasive radical hysterectomy (both total laparoscopic and total robotic radical hysterectomy) was associated with significantly worse disease-free survival and overall survival compared to open abdominal radical hysterectomy among women with early stage cervical cancer. Recurrence rates were also higher in the minimally invasive group.

This study aims to compare total laparoscopic radical hysterectomy and total abdominal radical hysterectomy in terms of disease-free survival and overall survival. Rates and characteristics of recurrence, incidence of complications and morbidity, impact on quality of life and cost-effectiveness will also be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed primary squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the uterine cervix
2. Patients with histologically confirmed stage IAI (+) LVSI, IA2, IB1, IB2 and IIA1 disease (TNM and 2018 FIGO staging for carcinoma of the uterine cervix)
3. Patients undergoing a Type II/Type III radical hysterectomy (Piver-Rutledge Classification) or Type B/Type C radical hysterectomy (Querleu-Morrow Classification)
4. Patients with adequate bone marrow, renal and hepatic function using Standard International Units 4.1 WBC > 3.0 x 109 cells/L 4.2 Platelets > 100 x 109 cells/L 4.3 Creatinine < 2.0 mg/dL 4.4 Bilirubin < 1.5 x upper normal limit and AST/SGOT or ALT/SGPT < 3 x upper normal limit
5. ECOG Performance Status of 0 or 1
6. Patients who have signed an approved Informed Consent
7. Patients with a prior malignancy if > 5 years ago with no current evidence of disease
8. Females aged 18 years or older
9. Negative serum pregnancy test ≤ 30 days of surgery in premenopausal women and women < 2 years after the onset of menopause

Exclusion Criteria:

1. Patients with any histology other than squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the uterine cervix
2. Stage IB3, IIA2-IV (TNM and 2018 FIGO staging for carcinoma of the uterine cervix)
3. Patients with evidence of metastatic disease by conventional imaging studies (CT Scan, MRI or PET CT Scan), enlarged pelvic or aortic lymph nodes > 2cm, or histologically positive lymph nodes
4. Patients with a history of pelvic or abdominal radiotherapy
5. Uterine size larger than 12 cm in length
6. Patients with contraindications to surgery or who are unfit for surgery with serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 820 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2031-07 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | 5 year
  the time from randomization to disease recurrence or death from cervical cancer
Overall Survival | 5 year
  the time from randomization to disease recurrence or death from any cause

SECONDARY OUTCOMES:
Recurrence Pattern | 5 years
  Recurrences will be described in detail and recorded according to date and location of first recurrence. The location can be designated as local, vault, pelvis or distal metastasis.
Intraoperative and Postoperative Complications | 1 year
  * Intraoperative complications - hemorrhage; injury to bladder, ureter, bowel; vascular injury; nerve injury
  * Perioperative complications (from post-surgery to discharge from hospital) - genitourinary (urinary tract infection, urinary retention), gastrointestinal (ileus), cardiac (myocardial infarction, atrial fibrillation), pulmonary (edema, atelectasis, pneumonia), renal and cerebrovascular morbidity. Wound and vault complications (infection, breakdown and dehiscence). Septicemia and thromboembolic complications (deep vein thrombosis and pulmonary embolism). Lymphocyst and abscess formation.
  * Early postoperative complications (<4 weeks from surgery): Wound and vault complications (infection, dehiscence). Urinary retention, urinary incontinence. Lymphocyst, lymphedema, abscess formation, or fistula formation.
  * Long term morbidity (4 weeks to 12 months from surgery): Urinary retention, urinary incontinence. lymphedema, incisional hernia formation, vaginal evisceration.
Impact on Quality of Life | 6 months
  Change in quality of life using Functional Assessment of Cancer Therapy Cervical (FACT-Cx) between baseline (pre-surgery) and 6 months after surgery. The FACT-CX comprises 42 items with 5 domains and a score range of 0-168.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Result] Wang YZ, Deng L, Xu HC, Zhang Y, Liang ZQ. Laparoscopy versus laparotomy for the management of early stage cervical cancer. BMC Cancer. 2015 Nov 24;15:928. doi: 10.1186/s12885-015-1818-4. PMID 26596955
- [Result] Shazly SA, Murad MH, Dowdy SC, Gostout BS, Famuyide AO. Robotic radical hysterectomy in early stage cervical cancer: A systematic review and meta-analysis. Gynecol Oncol. 2015 Aug;138(2):457-71. doi: 10.1016/j.ygyno.2015.06.009. Epub 2015 Jun 6. PMID 26056752
- [Result] Melamed A, Margul DJ, Chen L, Keating NL, Del Carmen MG, Yang J, Seagle BL, Alexander A, Barber EL, Rice LW, Wright JD, Kocherginsky M, Shahabi S, Rauh-Hain JA. Survival after Minimally Invasive Radical Hysterectomy for Early-Stage Cervical Cancer. N Engl J Med. 2018 Nov 15;379(20):1905-1914. doi: 10.1056/NEJMoa1804923. Epub 2018 Oct 31. PMID 30379613
- [Result] Ramirez PT, Frumovitz M, Pareja R, Lopez A, Vieira M, Ribeiro R, Buda A, Yan X, Shuzhong Y, Chetty N, Isla D, Tamura M, Zhu T, Robledo KP, Gebski V, Asher R, Behan V, Nicklin JL, Coleman RL, Obermair A. Minimally Invasive versus Abdominal Radical Hysterectomy for Cervical Cancer. N Engl J Med. 2018 Nov 15;379(20):1895-1904. doi: 10.1056/NEJMoa1806395. Epub 2018 Oct 31. PMID 30380365
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Bhatla N, Aoki D, Sharma DN, Sankaranarayanan R. Cancer of the cervix uteri. Int J Gynaecol Obstet. 2018 Oct;143 Suppl 2:22-36. doi: 10.1002/ijgo.12611. PMID 30306584
- [Result] Matsuo K, Machida H, Mandelbaum RS, Konishi I, Mikami M. Validation of the 2018 FIGO cervical cancer staging system. Gynecol Oncol. 2019 Jan;152(1):87-93. doi: 10.1016/j.ygyno.2018.10.026. Epub 2018 Oct 30. PMID 30389105
- [Result] Yan X, Li G, Shang H, Wang G, Han Y, Lin T, Zheng F. Twelve-year experience with laparoscopic radical hysterectomy and pelvic lymphadenectomy in cervical cancer. Gynecol Oncol. 2011 Mar;120(3):362-7. doi: 10.1016/j.ygyno.2010.11.033. Epub 2010 Dec 18. PMID 21168904
- [Result] Nam JH, Park JY, Kim DY, Kim JH, Kim YM, Kim YT. Laparoscopic versus open radical hysterectomy in early-stage cervical cancer: long-term survival outcomes in a matched cohort study. Ann Oncol. 2012 Apr;23(4):903-11. doi: 10.1093/annonc/mdr360. Epub 2011 Aug 12. PMID 21841155
- [Result] Yang L, Cai J, Dong W, Shen Y, Xiong Z, Wang H, Min J, Li G, Wang Z. Laparoscopic radical hysterectomy and pelvic lymphadenectomy can be routinely used for treatment of early-stage cervical cancer: a single-institute experience with 404 patients. J Minim Invasive Gynecol. 2015 Feb;22(2):199-204. doi: 10.1016/j.jmig.2014.09.009. Epub 2014 Oct 2. PMID 25281840
- [Result] Wang W, Chu HJ, Shang CL, Gong X, Liu TY, Zhao YH, Huang JM, Yao SZ. Long-Term Oncological Outcomes After Laparoscopic Versus Abdominal Radical Hysterectomy in Stage IA2 to IIA2 Cervical Cancer: A Matched Cohort Study. Int J Gynecol Cancer. 2016 Sep;26(7):1264-73. doi: 10.1097/IGC.0000000000000749. PMID 27643649
- [Result] Marcos-Sanmartin J, Lopez Fernandez JA, Sanchez-Paya J, Pinero-Sanchez OC, Roman-Sanchez MJ, Quijada-Cazorla MA, Candela-Hidalgo MA, Martinez-Escoriza JC. Does the Type of Surgical Approach and the Use of Uterine Manipulators Influence the Disease-Free Survival and Recurrence Rates in Early-Stage Endometrial Cancer? Int J Gynecol Cancer. 2016 Nov;26(9):1722-1726. doi: 10.1097/IGC.0000000000000808. PMID 27518143
- [Result] Uccella S, Bonzini M, Malzoni M, Fanfani F, Palomba S, Aletti G, Corrado G, Ceccaroni M, Seracchioli R, Shakir F, Ferrero A, Berretta R, Tinelli R, Vizza E, Roviglione G, Casarella L, Volpi E, Cicinelli E, Scambia G, Ghezzi F. The effect of a uterine manipulator on the recurrence and mortality of endometrial cancer: a multi-centric study by the Italian Society of Gynecological Endoscopy. Am J Obstet Gynecol. 2017 Jun;216(6):592.e1-592.e11. doi: 10.1016/j.ajog.2017.01.027. Epub 2017 Jan 29. PMID 28147240
- [Result] Piver MS, Rutledge F, Smith JP. Five classes of extended hysterectomy for women with cervical cancer. Obstet Gynecol. 1974 Aug;44(2):265-72. No abstract available. PMID 4417035
- [Result] Querleu D, Morrow CP. Classification of radical hysterectomy. Lancet Oncol. 2008 Mar;9(3):297-303. doi: 10.1016/S1470-2045(08)70074-3. PMID 18308255
- [Result] Sedlis A, Bundy BN, Rotman MZ, Lentz SS, Muderspach LI, Zaino RJ. A randomized trial of pelvic radiation therapy versus no further therapy in selected patients with stage IB carcinoma of the cervix after radical hysterectomy and pelvic lymphadenectomy: A Gynecologic Oncology Group Study. Gynecol Oncol. 1999 May;73(2):177-83. doi: 10.1006/gyno.1999.5387. PMID 10329031
- [Result] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Result] Lee CL, Wu KY, Huang KG, Lee PS, Yen CF. Long-term survival outcomes of laparoscopically assisted radical hysterectomy in treating early-stage cervical cancer. Am J Obstet Gynecol. 2010 Aug;203(2):165.e1-7. doi: 10.1016/j.ajog.2010.02.027. Epub 2010 May 11. PMID 20462565
- [Result] Lim TYK, Lin KKM, Wong WL, Aggarwal IM, Yam PKL. Surgical and Oncological Outcome of Total Laparoscopic Radical Hysterectomy versus Radical Abdominal Hysterectomy in Early Cervical Cancer in Singapore. Gynecol Minim Invasive Ther. 2019 Apr-Jun;8(2):53-58. doi: 10.4103/GMIT.GMIT_43_18. Epub 2019 Apr 29. PMID 31143623
- [Result] Lee CL. Minimally Invasive Therapy for Cancer: It is Time to Take Actions for Training System in Minimally Invasive Therapy After LACC Report. Gynecol Minim Invasive Ther. 2019 Jan-Mar;8(1):1-3. doi: 10.4103/GMIT.GMIT_132_18. Epub 2019 Jan 23. No abstract available. PMID 30783581